CLINICAL TRIAL: NCT01430351
Title: A Phase I Lead-In to a 2x2x2 Factorial Trial of Temozolomide, Memantine, Mefloquine, and Metformin as Post-Radiation Adjuvant Therapy of Glioblastoma Multiforme
Brief Title: Temozolomide, Memantine Hydrochloride, Mefloquine, and Metformin Hydrochloride in Treating Patients With Glioblastoma Multiforme After Radiation Therapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: <75 % participant accrual
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0374; NCI-2011-03038 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2011-0374 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2011-09-06; First posted 2011-09-08 (Estimated); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Glioblastoma; Gliosarcoma; Supratentorial Glioblastoma
MeSH Terms: conditions — Glioblastoma; Gliosarcoma | interventions — Mefloquine; Memantine; Metformin; Temozolomide

ARMS (8):
- Arm 1 (temozolomide) (Experimental): Patients receive temozolomide PO QD on days 1-5.
  Interventions: Drug: Temozolomide
- Arm 2 (temozolomide, memantine hydrochloride) (Experimental): Patients receive temozolomide PO as in Arm 1 and memantine hydrochloride PO BID.
  Interventions: Drug: Memantine Hydrochloride; Drug: Temozolomide
- Arm 3 (temozolomide, mefloquine) (Experimental): Patients receive temozolomide PO as in Arm 1 and 30 mg mefloquine PO QD on days 1-3 of week 1 and then days 2, 4, and 6 every other week.
  Interventions: Drug: Mefloquine; Drug: Temozolomide
- Arm 4 (temozolomide, metformin hydrochloride) (Experimental): Patients receive temozolomide PO as in Arm 1 and metformin hydrochloride PO BID.
  Interventions: Drug: Metformin Hydrochloride; Drug: Temozolomide
- Arm 5 (temozolomide, memantine hydrochloride, mefloquine) (Experimental): Patients receive temozolomide PO and memantine hydrochloride PO BID as in Arm 2, and mefloquine PO QD as in Arm 3.
  Interventions: Drug: Mefloquine; Drug: Memantine Hydrochloride; Drug: Temozolomide
- Arm 6 (temozolomide, memantine hydrochloride, metformin) (Experimental): Patients receive temozolomide PO and memantine hydrochloride PO BID as in Arm 2, and metformin hydrochloride PO BID as in Arm 4.
  Interventions: Drug: Memantine Hydrochloride; Drug: Metformin Hydrochloride; Drug: Temozolomide
- Arm 7 (temozolomide, mefloquine, metformin hydrochloride) (Experimental): Patients receive temozolomide PO as in Arm 1, mefloquine PO QD as in Arm 3, and metformin hydrochloride PO BID as in Arm 4.
  Interventions: Drug: Mefloquine; Drug: Metformin Hydrochloride; Drug: Temozolomide
- Arm 8 (TMZ, memantine hydrochloride, metformin, mefloquine) (Experimental): Patients receive temozolomide PO and memantine hydrochloride PO BID as in Arm 2, metformin hydrochloride PO BID as in Arm 4, and mefloquine PO QD as in Arm 3.
  Interventions: Drug: Mefloquine; Drug: Memantine Hydrochloride; Drug: Metformin Hydrochloride; Drug: Temozolomide

INTERVENTIONS:
Drug: Mefloquine — Given PO
  Arms: Arm 3 (temozolomide, mefloquine); Arm 5 (temozolomide, memantine hydrochloride, mefloquine); Arm 7 (temozolomide, mefloquine, metformin hydrochloride); Arm 8 (TMZ, memantine hydrochloride, metformin, mefloquine)
Drug: Memantine Hydrochloride — Given PO
  Other Names: Ebixia; Namenda
  Arms: Arm 2 (temozolomide, memantine hydrochloride); Arm 5 (temozolomide, memantine hydrochloride, mefloquine); Arm 6 (temozolomide, memantine hydrochloride, metformin); Arm 8 (TMZ, memantine hydrochloride, metformin, mefloquine)
Drug: Metformin Hydrochloride — Given PO
  Other Names: APO-Metformin; Cidophage; Dimefor; Glifage; Glucoformin; Glucophage; Glucophage ER; Metformin HCl; Riomet; Siofor
  Arms: Arm 4 (temozolomide, metformin hydrochloride); Arm 6 (temozolomide, memantine hydrochloride, metformin); Arm 7 (temozolomide, mefloquine, metformin hydrochloride); Arm 8 (TMZ, memantine hydrochloride, metformin, mefloquine)
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temcad; Temodal; Temodar; Temomedac

SUMMARY:
This phase I trial studies the side effects and best dose of combination chemotherapy in treating patients with glioblastoma multiforme after radiation therapy. Drugs used in chemotherapy, such as temozolomide, memantine hydrochloride, and metformin hydrochloride, work in different ways to stop the growth of tumor cells, either by killing them or stopping them from dividing. Mefloquine may help temozolomide, memantine hydrochloride, and metformin hydrochloride kill more cancer cells by making tumor cells more sensitive to the drug. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and tolerability of temozolomide (TMZ) in combination with metformin (metformin hydrochloride) (MFRMN) and/or mefloquine (MFLOQ) and/or memantine (memantine hydrochloride) (MEMTN) in patients receiving adjuvant therapy after completing external beam radiotherapy (XRT) in combination with chemotherapy for newly diagnosed glioblastoma multiforme (GBM).

SECONDARY OBJECTIVES:

I. To determine the median progression free survival (PFS); 6, 12, and 18 month PFS; and median overall survival (OS) in patients treated with temozolomide and a combination of metformin and/or mefloquine and/or memantine.

OUTLINE: This is a dose-escalation study. Patients are randomized to 1 of 8 different treatment arms.

ARM 1: Patients receive temozolomide orally (PO) once daily (QD) on days 1-5.

ARM 2: Patients receive temozolomide PO as in Arm 1 and memantine hydrochloride PO twice daily (BID).

ARM 3: Patients receive temozolomide PO as in Arm 1 and 30 mg mefloquine PO QD on days 1-3 of week 1 and then days 2, 4, and 6 every other week.

ARM 4: Patients receive temozolomide PO as in Arm 1 and metformin hydrochloride PO BID.

ARM 5: Patients receive temozolomide PO and memantine hydrochloride PO BID as in Arm 2, and mefloquine PO QD as in Arm 3.

ARM 6: Patients receive temozolomide PO and memantine hydrochloride PO BID as in Arm 2, and metformin hydrochloride PO BID as in Arm 4.

ARM 7: Patients receive temozolomide PO as in Arm 1, mefloquine PO QD as in Arm 3, and metformin hydrochloride PO BID as in Arm 4.

ARM 8: Patients receive temozolomide PO and memantine hydrochloride PO BID as in Arm 2, metformin hydrochloride PO BID as in Arm 4, and mefloquine PO QD as in Arm 3.

In all arms, courses repeat every 28 days for up to 24 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically proven supratentorial glioblastoma or gliosarcoma (World Health Organization [WHO] grade IV astrocytoma) will be eligible for this protocol; patients will be eligible if the original histology was low-grade glioma and a subsequent histological diagnosis of glioblastoma or gliosarcoma is made prior to any definitive treatment (radiotherapy, chemotherapy)
* All patients must sign an informed consent indicating that they are aware of the investigational nature of this study; patients must be registered prior to treatment with study drug
* Patients must have a Karnofsky performance status (KPS) of >= 60
* White blood cells (WBC) >= 3,000/ul (performed within 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1,500/mm^3 (performed within 14 days prior to registration)
* Platelet count of >= 100,000/mm^3 (performed within 14 days prior to registration)
* Hemoglobin >= 10 gm/dl (eligibility level for hemoglobin may be reached by transfusion) (performed within 14 days prior to registration)
* Serum glutamic oxaloacetic transaminase (SGOT) < 2 times upper limit of normal (ULN) (performed within 14 days prior to registration)
* Bilirubin < 2 times ULN (performed within 14 days prior to registration)
* Creatinine < 1.5 mg/dL (performed within 14 days prior to registration)
* For patients on mefloquine arm, a baseline electrocardiogram (EKG) without evidence of prolonged corrected QT (QTc) interval > 450 ms or clinically significant arrhythmia must be obtained within 14 days prior to registration
* A brain scan should be performed within 14 days prior to registration and steroid dosing should be stable or decreasing for at least 5 days; if the steroid dose is increased between the date of imaging and registration a new baseline magnetic resonance (MR)/computed tomography (CT) is required; the same type of scan, i.e., magnetic resonance imaging (MRI) or CT must be used throughout the period of protocol treatment for tumor measurement
* Patients must have completed standard radiation therapy with concurrent TMZ and must not have evidence of progressive disease on post treatment imaging
* Women of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin (B-HCG) pregnancy test documented within 72 hours of start of therapy
* Patients must be registered on the study within 5 weeks of completion of concurrent chemoradiation

Exclusion Criteria:

* Patients must not have any significant medical illnesses that, in the investigator's opinion, cannot be adequately controlled with appropriate therapy or would compromise the patient's ability to tolerate this therapy
* For mefloquine arm, patients with evidence of QTc interval > 450 ms or clinically significant arrhythmia on baseline EKG obtained within 14 days of registration will be ineligible for protocol enrollment
* Patients with a history of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission and off of all therapy for that disease for a minimum of 3 years, are ineligible
* Patients must not have active infection or serious intercurrent medical illness
* Patients must not be pregnant/breast feeding and must agree to practice adequate contraception (acceptable forms of birth control include condom with spermicide and/or diaphragm with spermicide, and non-barrier contraception such as tubal ligation, vasectomy, oral contraceptives, implanted levonorgestrel, vaginal hormonal contraceptive ring)
* Patients must not have any disease that will obscure toxicity or dangerously alter drug metabolism; patients with a history of psychosis/schizophrenia or cardiac disease requiring beta-blocker treatment (unable to change medication to non-beta blocker), anti-malarial drugs, or quinine or quinidine will not be eligible for enrollment to a mefloquine containing arm; patients who are on active treatment with one of the study drugs at the time of evaluation will not be eligible for enrollment to an arm containing that study drug
* For mefloquine arm, patients must not be on enzyme inducing anticonvulsants (EIAED); if the treating physician elects to change the medication to a non-enzyme inducing agent, a 2-week wash out period will be required after stopping EIAED prior to initiation of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2011-09-14 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Incidence of toxicities graded according to National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | During first 28 days

SECONDARY OUTCOMES:
Median progression free survival (PFS) | Up to 4 years
PFS | Up to 18 months
Median overall survival (OS) | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Vinay Puduvalli, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org